

#### **Informed Consent**

# INFORMED CONSENT/AUTHORIZATION FOR PARTICIPATION IN RESEARCH

Minimal Residual Disease Guided Maintenance Therapy with Belantamab Mafodotin and Lenalidomide After Autologous Hematopoietic Cell Transplantation in Patients with Newly Diagnosed Multiple Myeloma

| 2021-0201 | |
|---------------------------------------|-----------------------|
| Subtitle: GSK2857916 – ICF Model Safe | ty Language 23Jan2024 |
| Study Chair: Qaiser Bashir, I | MD |
| Participant's Name | Medical Record Number |

This is an informed consent and authorization form for a research study. It includes a summary about the study. A more detailed description of procedures and risks is provided after the summary.

This research has been reviewed and approved by an Institutional Review Board (IRB - a committee that reviews research studies).

#### STUDY SUMMARY

The goal of this clinical research study is to learn if belantamab mafodotin (BLENREP) can help to control multiple myeloma (MM) when given in combination with lenalidomide after a stem cell transplant. The study team will study this by measuring minimal residual disease (MRD). MRD refers to small numbers of cancer cells that remain in the body during or after treatment. The safety and tolerability of the study drug combination will also be studied.

This is an investigational study. Belantamab mafodotin was approved in the US in August 2020 under an FDA program called accelerated approval. In November 2022, belantamab mafodotin was removed from the market because a study done to confirm its ability to treat relapsed/refractory MM did not deliver a supporting result. However, the study did show that some patients may still benefit from treatment with belantamab mafodotin and that this benefit can be long lasting. It is your and your doctor's decision to take part in this study or to continue treatment if you are already enrolled in this study.

Lenalidomide is FDA approved and commercially available for the treatment of MM. It is considered investigational to study the effects of belantamab mafodotin in combination with lenalidomide in patients with MM who had had a stem cell transplant. The study doctor can explain how the study drug combination is designed to work.

This study also uses a test called clonoSEQ to measure MRD and will use the results to help make decisions about your treatment. clonoSEQ is FDA approved to measure MRD, but it is not approved for use related to treatment decisions.

The study drug combination may help prevent MM from coming back. Future patients may benefit from what is learned. There may be no benefits for you in this study.

Your participation is completely voluntary. Before choosing to take part in this study, you should discuss with the study team any concerns you may have, including side effects, potential expenses, and time commitment.

You can read a list of potential side effects below in the Possible Risks section of this consent.

You may take the study drugs for as long as the study doctor thinks it is in your best interest.

Belantamab mafodotin will be provided at no cost to you while you are on study. You and/or your insurance provider will be responsible for the cost of lenalidomide and all tests and procedures performed in this study.

You may choose not to take part in this study. Instead of taking part in this study, you may choose to receive the standard treatment for the disease. The study doctor will discuss the standard treatments available to you. You may choose to receive other investigational therapy, if available. The study doctor will discuss the possible risks and benefits of these treatments. You may choose not to receive treatment for cancer at all. In all cases, you will receive appropriate medical care, including treatment for pain and other symptoms of cancer.

#### 1. STUDY DETAILS

#### **Screening Tests**

Signing this consent form does not mean that you will be able to take part in this study. The following screening tests will help the doctor decide if you are eligible:

- You will have a physical exam.
- You will have an eye exam performed by an eye doctor.
- Blood (about 3 tablespoons) will be drawn for routine tests, immune system
  testing, viral testing (to check for viruses like hepatitis B/C and HIV [the AIDS
  virus]), and tests to check the status of the disease.

- You will have a bone marrow biopsy and aspirate to check the status of the
  disease and for cytogenetic testing. Cytogenetic testing looks at how genetic
  changes to cells may affect how the disease may react to the study drug. To
  collect a bone marrow aspirate and biopsy, an area of the hip or other site is
  numbed with anesthetic, and a small amount of bone marrow and/or bone is
  withdrawn through a large needle.
- You will have an EKG and an echocardiogram (ECHO) to check your heart function.
- You will have a PET scan to check the status of the disease. If the study doctor thinks it is needed, you may have additional imaging scans such as a bone survey, CT scan, MRI, or PET-CT scan. A bone survey is a series of xrays of all or most of the bones in your body.
- Urine will be collected for routine tests and to check the status of the disease.
   You will be asked to collect your urine over 24 hours for these tests. The study team will give you a container and instructions on how to collect the urine.
- If you can become pregnant, a blood sample will be used for a pregnancy test within 10-14 days and 24 hours before your first dose of lenalidomide. To take part in this study, you must not be pregnant.

If needed, some of these tests may need to be repeated during screening. The study team will let you know if this is needed.

The study doctor will discuss the screening test results with you. If the screening tests show that you are not eligible to take part in this study, you will not be enrolled. Other treatment options will be discussed with you.

Up to 94 participants will be enrolled in this study. All will take part at MD Anderson.

#### **Study Drug Administration**

You are scheduled to have a stem cell transplant as part of your standard of care. You will sign a separate consent form describing the stem cell transplant, including its risks. **About 60-180 days after your stem cell transplant**, you will start to receive the study drugs.

The study drugs will be given to you in cycles. Each cycle will last 84 days for a maximum of 12 cycles.

You will receive belantamab mafodotin by vein over about 30 minutes on **Day 1 of each cycle**.

You will also take lenalidomide by mouth **every day of each cycle.** You should take lenalidomide with a glass (about 8 ounces) of water at about the same time each day. You may take lenalidomide with or without food. Swallow the capsule whole; do not break open or chew the capsule. If you miss a dose and it has been less than 12 hours since the usual dosing time, you should take the missed dose. However, if you miss a dose and it has been more than 12 hours since the usual dosing time, you

should not make up the missed dose. Wait and take the next dose as scheduled. Do not take 2 doses to make up for a missed dose.

If the study doctor thinks it is needed, your dose level of belantamab mafodotin and/or lenalidomide may be changed. This will be discussed with you.

If a dose of belantamab is delayed due to side effects, your doctor may decide if it is in your best interest to wait for 6-12 weeks before giving you your next dose.

You may be given standard drugs during this study to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

You will no longer be able to receive the study drugs if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

### **Study Visits**

# On Day 1 of each cycle:

- You will have a physical exam.
- You will have an eye exam performed by an eye doctor within 5 days before your belantamab mafodotin dose.
- Blood (about 3 teaspoons) will be drawn for routine tests, immune system testing, and tests to check the status of the disease.
- Urine will be collected for routine tests and to check the status of the disease. You will need to collect your urine over 24 hours for these tests. The study staff will give you a container and instructions on how to collect the urine.

# At Week 4 of every Cycle:

- You will have a physical exam. This may be performed virtually (for example, by video call) if needed.
- Blood (about 3 tablespoons) will be drawn for routine tests, immune system
  testing, and tests to check the status of the disease. If it is more convenient
  for you, you may have some of these blood tests done at a local lab or
  doctor's office that is closer to your home. In some cases, some blood tests
  may not need to be performed (based on the doctor's discretion). This will be
  discussed with you.

# At Week 8 of every Cycle:

 You will have a physical exam. This may be performed virtually (for example, by video call) if needed. Blood (about 3 tablespoons) will be drawn for routine tests, immune system
testing, and tests to check the status of the disease. If it is more convenient
for you, you may have some of these blood tests done at a local lab or
doctor's office that is closer to your home. In some cases, some blood tests
may not need to be performed (based on the doctor's discretion). This will be
discussed with you.

### About 1, 2, and 3 years after your first dose:

- You will have a bone marrow biopsy to check the status of the disease and for cytogenetic testing.
- You will have a PET scan to check the status of the disease.

# If the disease gets worse, the following tests will also be performed:

- You will have a bone marrow biopsy to check the status of the disease and for cytogenetic testing.
- Blood (about 3 teaspoons) will be drawn for routine tests, immune system tests, and tests to check the status of the disease.
- Urine will be collected to check the status of the disease. You will need to collect your urine over 24 hours for these tests.
- You will have a PET scan to check the status of the disease.

At any time the study doctor thinks it is needed, the above listed tests and procedures may be repeated to check on your health. You may also have CT scans, MRIs, or bone surveys to check the status of the disease.

# **Follow-Up Visit**

**About 70 days after you stop taking the study drugs**, you will have a follow-up visit. The following tests and procedures will be performed at this visit:

- You will have a physical exam.
- You will have an eye exam performed by an eye doctor.
- Blood (about 3 teaspoons) will be drawn for routine tests.
- You will have a bone marrow biopsy to check the status of the disease and for cytogenetic testing.

You will have eye exams by an eye doctor every 3 months for up to 1 year after stopping study treatment, unless the eye doctor thinks it is no longer needed.

#### **Pregnancy Tests**

If you can become pregnant, you will also have blood and/or urine pregnancy tests throughout study treatment at the following time points:

- One (1) time a week during the first 4 weeks of lenalidomide treatment, then ever 4 weeks (if you have regular menstrual periods) or 2 weeks (if you have irregular menstrual periods) after that
- As soon as possible after stopping lenalidomide treatment and then again about 28 days later; if you have irregular menstrual periods, you will have an additional test about 14 days after stopping lenalidomide treatment

• About 70 days and 4 months after stopping belantamab mafodotin treatment

#### Other Information

Belantamab mafodotin may cause eye irritation. To help treat or prevent eye irritation during this study, the follow precautions will be taken:

- You may use cooling eye masks at start of each belantamab infusion and for up to 4 hours afterwards, as tolerated and needed.
- Starting with your first belantamab mafodotin infusion, you will use artificial tears (eye drops) in each eye at least 4-8 times every day until you stop taking belantamab mafodotin.
- You cannot wear contact lenses during this study. If the eye doctor thinks it is safe for you to do so, you may restart wearing contact lenses after you stop taking belantamab mafodotin.

#### 2. POSSIBLE RISKS

While on this study, you are at risk for side effects. You should discuss these with the study doctor. The more commonly occurring side effects are listed in this form, as are rare but serious side effects. You may also want to ask about uncommon side effects that have been observed in small numbers of patients but are not listed in this form. Many side effects go away shortly after treatment is stopped, but in some cases side effects may be serious, long-lasting or permanent, and may even result in hospitalization and/or death.

Side effects will vary from person to person, and some may occur after you have stopped receiving treatment. Tell the study staff about any side effects you may have, even if you do not think they are related to the study drugs/procedures.

Belantamab mafodotin and lenalidomide may each cause low blood cell counts (red blood cells, white blood cells, and/or platelets):

- A low red blood cell count (anemia) may cause difficulty breathing and/or fatigue. You may need a blood transfusion.
- A low white blood cell count increases your risk of infection (such as pneumonia and/or severe blood infection). Infections may occur anywhere and become life-threatening. Symptoms of infection may include fever, pain, redness, and difficulty breathing. If you have a fever, please contact your study doctor.
- A low platelet count increases your risk of bleeding (such as nosebleeds, bruising, stroke, and/or digestive system bleeding). Bleeding may be serious or life threatening and you may need a platelet transfusion.

#### **Belantamab Mafodotin Side Effects**

Belantamab mafodotin is an approved drug in the European Union, United Kingdom, Switzerland, Singapore, Hong Kong and Israel with ongoing clinical development; therefore, not all of its side effects are known at this time. As of 27 February 2024,

over 1700 people worldwide with multiple myeloma have received belantamab mafodotin across all ongoing and completed clinical studies.

Some common side effects reported with belantamab mafodotin are described below:

# **Eye Problems**

Some people who have received belantamab mafodotin in clinical studies developed problems in the front part of the eye called the cornea. Sometimes the changes can only be observed by an eye care specialist during eye examination, and they do not result in any symptoms. Those changes might be more frequent in patients who had problems with dry eye before treatment with belantamab mafodotin. However, some patients develop symptoms related to belantamab mafodotin. The symptoms could range from a feeling of dryness in the eye to more severe symptoms, like blurry vision or changes in your eyesight that could affect your ability to see things clearly and may affect your reading ability or lead to difficulty in driving.

These effects typically go away if the study drug is paused and the dose reduced upon re-start, but please discuss with your study doctor if you have questions. In severe cases, sores can develop on the eye, possibly with infection. Even if treated, this could potentially lead to scarring which may permanently affect your eyesight including severe vision loss.

If you experience new eye symptoms (such as pain or irritation, blurry vision, or feeling like something is in your eye), you should urgently seek medical attention by an eye care specialist. Your eyes will be examined repeatedly during the study, as it is important to monitor the effects of belantamab mafodotin on your eyes.

If you develop problems with your eyesight or other problems with your eyes, do not drive or operate heavy machinery until you have had your eyes examined by an eye care specialist.

#### Abnormal bruising and bleeding

Belantamab mafodotin can decrease the number of blood cells called platelets, which help to clot your blood. Symptoms of low platelet counts (called thrombocytopenia) can include abnormal bruising of your skin, bleeding for longer than usual after your blood has been drawn, or bleeding from your nose or gums. In some cases, the bleeding can occur from other areas of your body. Bleeding may be serious or life-threatening and may require a transfusion. Your study doctor will closely monitor your platelets by checking your blood tests before you start your treatment and regularly during the study.

#### Infusion-related reactions

Some people may have allergic-like reactions when they receive an infusion of belantamab mafodotin. These usually develop within minutes or hours but can develop up to 24 hours after your dose is given. It is a reaction to the drug being a foreign protein, and you may have flushing, chills, fever, problems with breathing,

feeling like your heart is racing, or a drop in blood pressure (which may cause you to feel dizzy, light-headed, or like you're going to faint). You will usually spend an hour after your dose to check whether you will develop these symptoms but if you experience any of these symptoms at any time contact your study doctor immediately.

# Inflammation of the lungs

Some people who have received belantamab mafodotin experienced inflammation of the lungs which can cause cough, shortness of breath, and difficulty breathing and in rare cases, death. It is not certain if belantamab mafodotin causes the inflammation or not. If you experience new or worsening breathing problems like cough or shortness of breath with an unknown cause, contact your study doctor immediately.

### Excess protein in the urine

Some people receiving belantamab mafodotin have developed excess levels of protein (called albumin) in the urine, which can sometimes be a sign of a kidney disorder.

Your study doctor will closely monitor protein levels in your urine regularly during the study. If your urine looks foamy or frothy or if you notice new swelling or more swelling than usual in your feet, legs, or other parts of your body, contact your study doctor immediately.

#### Side effects

The side effects described below are from 95 people with relapsed/refractory multiple myeloma who received at least 1 dose of belantamab mafodotin in 1 study, at a dose of 2.5 mg/kg.

# The most common side effects occurring in more than 10% of participants (10 or more out of 100 participants) were:

- Eye side effects: blurred vision, dry/itchy eyes, changes in vision, eye discomfort, difficulty seeing at night, swelling, or other changes to the front part of eye
- Low number of blood cells called platelets, which may cause bleeding and easy bruising; bleeding may be serious or life-threatening and may require a transfusion
- Anemia (when your body has fewer red blood cells than normal)
- Feeling sick to your stomach (nausea)
- Feeling tired (fatigue)
- Abnormal liver tests
- Fever (if you have a fever, please contact your study doctor)
- Pneumonia, or other lung infections
- Cold or cold-like symptoms (upper respiratory tract infection)
- Low number of certain types of white blood cells called neutrophils (neutropenia) and lymphocytes (lymphopenia), which could increase the risk of infection; if you have a fever, please contact your study doctor immediately
- Diarrhea

 Reactions from the infusion of belantamab mafodotin, usually happening within the first 24 hours after the infusion: symptoms may include: flushing, chills, fever, difficulty breathing, rapid heartbeat, or a drop in blood pressure (feeling light-headed)

Other common side effects seen in 1% to 10% of participants (between 1 to 10 out of 100 participants) were:

- Other eye side effects: eye irritation, abnormal sensitivity of the eyes to light, and sores on the eyes possibly with infection.
- Increased albumin, a type of protein, in the urine (albuminuria)
- An increase in an enzyme released into the blood when muscle is damaged (creatine phosphokinase)
- Vomiting

In another study which is testing belantamab mafodotin in combination with 2 medicines already approved for the treatment of relapsed refractory multiple myeloma (called lenalidomide and dexamethasone), 2 patients who had low white blood cell (neutrophil) counts developed serious infections which led to death.

If you have fever at any point while you are in this study, contact your study doctor immediately.

**Embryo-fetal toxicity**: Belantamab mafodotin may harm an unborn baby. You must have negative pregnancy tests to continue in the study if you are a woman who can have children. See section called "**Pregnancy Related Risks**" below for further details.

**Fertility**: Belantamab mafodotin treatment may affect men and women's ability to have children. See section called "**Pregnancy Related Risks**" below for further details.

There may be other side effects that may happen that are not known now. For example, all drugs can cause an allergic reaction in some patients. Certain problems can become worse if not treated quickly. Call the study doctor right away if:

- You feel very tired or faint
- You feel pain or sick in your stomach and you do not want to eat
- You bruise easily or develop itching
- You have yellow eyes or skin, or dark urine
- You become confused

#### **Lenalidomide Side Effects**

Common (occurring in more than 20% of patients)

- swelling (arm/leg)
- fatigue
- fever
- dizziness
- skin rash/itching
- inflammation of the stomach and/or intestines
- diarrhea/constipation
- nausea
- low blood cell counts (red, platelets, white)
- muscle cramps/spasms
- weakness
- pain
- lung inflammation
- cough
- infection (including upper respiratory tract, nose, sinuses, and/or throat)

# Occasional (occurring in 3-20% of patients)

- swelling
- high blood pressure
- low blood pressure (possible dizziness/ fainting)
- chest pain (possibly due to heart trouble)
- irregular heartbeat
- blood clots in a vein (possible pain, swelling, and/or redness)
- chills/shivering
- headache
- difficulty sleeping
- abnormal sensation (such as pins and needles)
- abnormal salts, minerals, and/or acids in the blood (possible weakness, swelling, fatigue, low blood pressure, organ failure, heart problems, changes in mental status, and/or seizure)

- sweating
- skin redness
- dry skin
- underactive thyroid gland (possible weight gain, heart failure, and/or constipation)
- abnormal taste
- dry mouth
- dehydration
- vomiting
- weight loss
- loss of appetite
- abdominal pain
- difficult and/or painful urination
- increased risk of bleeding
- numbness
- nerve damage (possible loss of motor or sensory function)
- abnormal liver tests (possible liver damage)

- kidney failure
- kidney stones
- runny nose
- blockage in the lung (possible pain, shortness of breath, and/or failure to breathe)
- build-up of fluid around the lungs
- flu-like illness
- nosebleed
- sore throat
- pain and/or inflammation at the tumor site
- allergic reaction
- breakdown products of the cancer cells entering the blood stream (possible weakness, low blood pressure, muscle cramps, kidney damage, and/or other organ damage)

Lenalidomide may occasionally cause you to develop another type of cancer (such as leukemia [blood cancer], lymphoma [cancer of the lymph nodes], skin cancer, lung cancer, prostate cancer, or other solid tumors).

Rare but serious (occurring in fewer than 3% of patients)

- tissue swelling
- stroke
- very severe blistering skin disease (with ulcers of the skin and digestive tract)
- very severe blistering skin disease (loss of large portion of skin)
- skin rash (possible fever/lymph node swelling/inflammation of internal organs/abnormal blood cell counts)
- overactive thyroid gland (possible weight loss, heart rate changes, and/or sweating)

- low blood levels of sodium (possible headache, confusion, seizures, and/or coma)
- inflammation of the bile tract (possible blockage)
- abnormal blood test (possible heart problems)
- bacteria in the blood
- liver damage
- reactivation of hepatitis
   B infection (possible liver damage) and/or herpes zoster
- abnormal liver tests (possible yellowing of the skin and/or eyes)

- low oxygen level in the blood (possible lightheadedness)
- severe life-threatening infection (possible low blood pressure, kidney failure, and/or heart failure)
- graft-versus-host disease (when transplanted donor tissue attacks the tissues of the recipient's body)
- organ transplant rejection

Lenalidomide may rarely cause problems with collecting your own stem cells which may cause you to be unable to receive certain types of stem cell transplants.

# It is not known how often the following side effects may occur:

- fast/slow heartbeat
- heart failure or other severe heart problems
- shock (possibly caused by heart damage)
- heart attack
- decreased supply of blood to a body part (such as the heart)
- enlarged heart
- bleeding around the brain
- abnormal blood clotting
- difficulty forming or speaking words
- migraine
- temporary stroke symptoms
- confusion
- depression

- inflammation of the colon (possible abdominal pain and/or diarrhea)
- digestive system bleeding
- difficulty swallowing
- chronic heartburn and indigestion
- intestinal blockage
- hole in the intestines (possibly leaking contents into the abdomen)
- decreased blood flow to part of the bowel or other body part (possibly causing tissue death)
- bleeding or blood in stool

- blockage of the bile tract (possible body yellowing and/or abdominal pain)
- difficulty walking
- falling
- painful joint inflammation
- pelvic pain
- broken bones (such as leg, pelvis, hip, rib, collapsed spine bones)
- build-up of bone-like crystals (calcium phosphate) in different parts of the body (possible pain and/or decreased organ function)
- build-up of bodily waste products in the blood

- loss of alertness
- skin condition with fever and skin lesions
- skin bump
- immune response that causes an overactive thyroid gland (possible fast heartbeat, sweating, weight loss, nervousness, and/or eye bulging)
- low blood sugar
- inflammation of the pancreas (possible abdominal pain)

- pockets of pus in or near the anus
- death of spleen tissue
- gallbladder inflammation (possible abdominal pain)
- tarry stool
- blood in the urine
- destruction of red blood cells (possible anemia)
- bleeding after procedures
- liver failure

- (possible kidney damage)
- kidney damage
- abnormal kidney tests (possible kidney damage)
- abnormal growth in the kidneys
- difficulty breathing, possibly due to lung damage or fluid in the lung
- wheezing
- worsening of disease

**Using the study drugs together** may cause side effects that are not seen when each is given alone. The study drug combination may also increase the frequency and/or severity of the side effects listed above.

### **Other Risks**

**Blood draws** may cause pain, bleeding, and/or bruising. You may faint and/or develop an infection with redness and irritation of the vein at the site where blood is drawn. Frequent blood collection may cause anemia (low red blood cell count), which may create a need for blood transfusions.

Having **bone marrow biopsies/aspirates** performed may cause pain, bruising, bleeding, redness, low blood pressure, swelling, and/or infection at the site of the biopsies. An allergic reaction to the anesthetic may occur. A scar may form at the biopsy site.

**X-rays** send a small amount of radiation though the body. All radiation adds up over a lifetime and may increase the risk of a new cancer forming.

**EKGs and ECHOs** may cause discomfort while lying on the exam table, and the tape on the EKG pads may cause skin irritation.

**MUGA scans** may cause allergic reactions to the radioactive tracer, injection site soreness, and/or swelling. They may cause damage to cells or tissue from being exposed to the radiation used in the scan. These side effects may occur in less than 10% of patients.

During the **MRI**, you may feel mild vibrations throughout your body. The machine will produce a loud knocking noise. This is normal. You will be given earplugs to protect your ears. Some people, especially those who tend to feel uncomfortable in small or

closed spaces, may feel "closed in" and become anxious while in the scanner. The scanner has an intercom, which will allow you to speak to the staff during the procedure. If you feel ill or anxious during scanning, tell the MRI staff and the scanning will be stopped if you wish. The MRI will require a catheter to be inserted into one of your veins in order to inject the MRI contrast agent. This may cause skin irritation, bleeding, and/or infection. You may have an allergic reaction to the contrast agent.

The magnetic field used in MRI scanning may harm you if you have certain types of metal in your body (as might be found in pacemakers, neurostimulators, or certain clips). It may cause problems with devices, such as pacemakers. If you have metal in your body or devices such as a pacemaker, you should discuss this with the study doctor.

**CT scans** send x-rays through the body at many different angles. You will be exposed to a small dose of radiation. All radiation adds up over a lifetime and may increase the risk of new cancer forming. Some people may feel "closed in" while lying in the scanner. However, the scanner is open at both ends, and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or radiology technicians will give comfort, or the scanning will be stopped. Solution may also be given by vein to make the x-ray pictures more accurate. This may cause an uncomfortable feeling of warmth, nausea, and/or severe allergic reactions. The solution injection may also cause pain, bleeding, bruising, hives, and/or itching.

A **PET scan** may cause you to feel "closed in" while lying in the scanner. However, the scanner is open at both ends and an intercom allows you to talk with doctors and staff. If you feel ill or anxious during scanning, doctors and/or technicians will give comfort or the scanning will be stopped.

The PET scan exposes your body to radiation. The radioactive solution does not remain in your system for a long period of time. However, you should wait 2 hours before holding an infant or getting close to a pregnant woman to avoid exposing them to radiation. You should drink fluids after the scan to help remove the solution from your system.

During the **eye exam**, your pupils will be dilated with eye drops to allow a good view of the back of the eye. This will result in some blurred vision lasting for a few hours. You will not be able to drive during this time.

Although every effort will be made to keep study data safe, there is a chance that your personal health information could be lost or stolen, which may result in a **loss of confidentiality**. All study data will be stored in password-protected computers and/or locked file cabinets and will continue to be stored securely after the study.

This study may involve unpredictable risks to the participants.

## **Pregnancy Related Risks**

Taking part in this study can result in risks to an unborn or breastfeeding baby, so you should not become pregnant, breastfeed a baby, or father a child while on this study. You must use birth control during the study if you are sexually active. Belantamab mafodotin may also affect your ability to have children in the future. If you may want to have children in the future, you should consider freezing and storing your eggs/sperm before beginning the study treatment. Talk to the study doctor if you have questions about this process.

Birth Control Specifications: If you can become pregnant, you must use a highly effective birth control method plus 1 additional method during this study and for 28 days after your last dose of lenalidomide or 4 months after your last dose of belantamab mafodotin, whichever is longer:

- Highly effective methods include:
  - Combined (estrogen- and progestogen-containing) hormonal birth control associated with stopping ovulation (such as birth control pills, intravaginal ring, patches, or injections)
  - Progestogen-only birth control hormonal birth control associated with stopping ovulation (such as birth control pills, injections, or implant)
  - Intrauterine device (IUD) or intrauterine hormone-releasing system (IUS)
  - Bilateral tuba occlusion ("tubes tied")
  - Vasectomy of yourself or your sale male partner
- Additional methods include:
  - Latex condoms
  - Diaphragm
  - Cervical cap

If you can father a child, you must use condoms, even if you have had a successful vasectomy, during this study and for 28 days after your last dose of lenalidomide or 6 months after your last dose of belantamab mafodotin, whichever is longer.

Males: Do not donate sperm during this study and for 4 weeks after your last dose of lenalidomide and for 6 months after your last dose of belantamab mafodotin. Tell the doctor right away if your partner becomes pregnant or suspects pregnancy. If your partner/spouse becomes pregnant while you are on this study, the study supporter (GlaxoSmithKline, Inc.) would like to collect information about the pregnancy. The study supporter will make their contact information available to you so that, if you and your partner wish to, you can share information about the outcome of the pregnancy with the study supporter. If you and/or your partner choose not to share this information, it will not result in any penalty or loss of benefits to which you are otherwise entitled.

Females: Do not donate eggs (ova, oocytes) during this study and for 4 weeks after your last dose of lenalidomide or 4 months after your last dose of belantamab mafodotin, whichever is longer. If you are pregnant, you will not be enrolled on this

study. If you become pregnant or suspect that you are pregnant, you must tell your doctor right away. The study supporter will ask for information about the pregnancy. You will be followed up for up to 6 - 8 weeks after the estimated delivery date to check on how your delivery went and the health of your baby.

Mothers must not breastfeed a baby while on this study and for 4 months after the last dose of study drug.

Getting pregnant will result in your removal from this study.

There are additional risks associated with lenalidomide. If lenalidomide is taken during pregnancy, it may cause birth defects or death to an unborn baby. Because of this risk, all patients taking lenalidomide must read the following statements that apply to them according to gender and menopausal status.

#### FOR FEMALES WHO ARE ABLE TO BECOME PREGNANT\*

TIME.

\*(Sexually mature female who: 1) has not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or 2) has not been naturally postmenopausal for at least 24 consecutive months)

Please read thoroughly and initial each space provided if you understand each statement

\_\_\_\_\_: I understand that birth defects may occur with the use of lenalidomide. I have been warned by my doctor that my unborn baby may have birth defects and can even die, if I am pregnant or become pregnant while I am taking lenalidomide.
\_\_\_\_: I understand that I must NOT take lenalidomide if I am pregnant, breast-feeding a baby or able to get pregnant and not using 2 reliable methods of birth control.
\_\_\_\_\_: If I am having sexual relations with a man, my uterus and/or both ovaries have not been removed, I have had at least one menstrual period in the past 24 months and/or my menses stopped due to treatment of my disease, I understand that I am able to become pregnant. I must use one highly effective method of birth control plus one additional effective method of birth control (contraception) at the SAME

Highly Effective Methods
Intrauterine device (IUD)
Hormonal (birth control pills, injections, implants)
Tubal ligation
Partner's vasectomy

Additional Effective Methods
Latex condom
Diaphragm
Cervical Cap

\_\_\_\_\_: These birth control methods must be used during the following time periods related to this study: 1) for at least 28 days before starting lenalidomide therapy; 2) while participating in the study; during interruptions in therapy and 3) for at least 28 days after lenalidomide has been stopped. I must use these methods unless I completely abstain from heterosexual sexual contact. If a hormone (birth control pill, injection, patch, or implant) or IUD method is not medically possible for me, I may use another highly effective method or two barrier methods AT THE SAME TIME.

| and 24 hours prior to starting lenalidomide therapy, even if I have not had my menses due to treatment of my disease or had as little as one menstrual period in the past 24 months. If I have regular or no menstrual cycles, I will then have pregnancy tests every week for the first 28 days, then every 28 days while I am taking lenalidomide, again when I have been taken off of lenalidomide therapy and then 28 days after I have stopped taking lenalidomide. If I have irregular menstrual cycles, I will have pregnancy tests every week for the first 28 days, then every 14 days while I am taking lenalidomide, again when I have been taken off of lenalidomide therapy, and then 14 days and 28 days after I have stopped taking lenalidomide. |
|---|
| : I know I must immediately stop taking lenalidomide and inform my doctor, if I become pregnant while taking the drug, if I miss my menstrual period or have unusual menstrual bleeding, if I stop using 2 reliable forms of birth control, or if I think for any reason that I may be pregnant. I must talk to my doctor before changing any birth control methods. |
| : I am not now pregnant, nor will I try to become pregnant for at least 28 days after I have completely finished taking lenalidomide. : I understand that lenalidomide will be prescribed only for me. I must not share it with ANYONE, even someone that has similar symptoms to mine. It must be |
| kept out of reach of children and should never be given to females who are pregnant or able to have children. : I agree any unused drug supply will be returned to the research site at each visit. |
| : I know that I cannot donate blood while taking lenalidomide and for 28 days after stopping lenalidomide. Study patients who become pregnant will be monitored throughout the pregnancy and will continue to be monitored for 30 days after delivery (premature delivery, aborted fetus, full-term pregnancy, or no longer pregnant). |
| FOR ALL MALES Please read thoroughly and initial each space provided if you understand each statement: |
| : I understand that birth defects may occur with the use of lenalidomide. I have been warned by my doctor that an unborn baby may have birth defects and can ever die, if a female is pregnant or becomes pregnant while taking lenalidomide: I have been told by my doctor that I must NEVER have unprotected sexual contact with a female who can become pregnant. Because it is known that lenalidomide is present in semen, my doctor has explained that I must completely abstain from sexual contact with females who are pregnant or able to become pregnant, or I must use a latex condom every time I engage in any sexual contact with females who are pregnant or may become pregnant. I must do this while I am taking lenalidomide and for 28 days after I stop taking lenalidomide, even if I have had a successful vasectomy. |
| : I know I must inform my doctor if I have unprotected sexual contact with a female who is pregnant or can become pregnant or if I think, for ANY REASON, that my sexual partner may be pregnant. Female partners of male patients taking |

\_\_\_\_: I know I must have a pregnancy test done by my doctor within 10 – 14 days

| pregnant. |
|---|
| : I understand that lenalidomide will be prescribed only for me. I must not share it with ANYONE, even someone that has similar symptoms to mine. It must be kept out of reach of children and should never be given to females who are able to |
| have children. |
| : I agree any unused drug supply will be returned to the research site at each visit. |
| : I know that I cannot donate blood, sperm, or semen while taking lenalidomide and for 28 days after stopping lenalidomide. |
| FOR FEMALES WHO ARE NOT ABLE TO BECOME PREGNANT Please read thoroughly and initial each space provided if you understand each statement. |
| : I understand that birth defects may occur with the use of lenalidomide. I have been warned by my doctor that an unborn baby may have birth defects and can even die, if a female is pregnant or becomes pregnant while taking lenalidomide: I certify that I am not now pregnant, nor am I of child bearing potential as I have been in a natural menopause for at least 24 months (been through the change in life without even 1 menstrual period for the past 24 months); or I had my uterus |
| removed (hysterectomy) or had both my ovaries removed (bilateral oophorectomy). : I understand that lenalidomide will be prescribed only for me. I must not share it with ANYONE, even someone that has similar symptoms to mine. It must be kept out of reach of children and should never be given to females who are pregnant or able to have children. |
| : I agree any unused drug supply will be returned to the research site at each visit. |
| : I know that I cannot donate blood while taking lenalidomide and for 28 days after stopping lenalidomide. |
| ALL PATIENTS |
| You will be counseled at least every 28 days about not sharing lenalidomide (and |

lenalidomide should be advised to call their own physician immediately if they get

other study drugs), the potential risks of fetal exposure, abstaining from blood and other donations, the risk of changes in blood counts and blood clots, and you will be reminded not to break, chew or open lenalidomide capsules. You will be provided with the "Lenalidomide Information Sheet for Patients Enrolled in Clinical Research Studies" with each new supply of lenalidomide as a reminder of these safety issues. You must receive counseling and complete phone surveys as required by the Revlimid REMS program.

Pregnant females or females that are able to become pregnant should not handle or administer lenalidomide unless they are wearing gloves.

#### 3. COSTS AND COMPENSATION

If you suffer injury as a direct result of taking part in this study, MD Anderson health providers will provide medical care. However, this medical care will be billed to your insurance provider or you in the ordinary manner. You will not be reimbursed for expenses or compensated financially by MD Anderson or GlaxoSmithKline, Inc. for this injury. You may also contact the Chair of MD Anderson's IRB at 713-792-6477 with questions about study-related injuries. By signing this consent form, you are not giving up any of your legal rights.

Certain tests, procedures, and/or drugs that you may receive as part of this study may be without cost to you because they are for research purposes only. However, your insurance provider and/or you may be financially responsible for the cost of care and treatment of any complications resulting from the research tests, procedures, and/or drugs. Standard medical care that you receive under this research study will be billed to your insurance provider and/or you in the ordinary manner. Before taking part in this study, you may ask about which parts of the research-related care may be provided without charge, which costs your insurance provider may pay for, and which costs may be your responsibility. You may ask that a financial counselor be made available to you to talk about the costs of this study.

Samples that are collected from you in this study may be used for the development of treatments, devices, new drugs, or patentable procedures that may result in commercial profit.

There are no plans to compensate you for any patents or discoveries that may result from your participation in this research.

You will receive no compensation for taking part in this study.

#### **Additional Information**

- 4. You may ask the study chair (Dr. Qaiser Bashir, at 713-792-8750) any questions you have about this study. You may also contact the Chair of MD Anderson's Institutional Review Board (IRB a committee that reviews research studies) at 713-792-6477 with any questions that have to do with this study or your rights as a study participant.
- 5. You may choose not to take part in this study without any penalty or loss of benefits to which you are otherwise entitled. You may also withdraw from participation in this study at any time without any penalty or loss of benefits. If you decide you want to stop taking part in the study, it is recommended for your safety that you first talk to your doctor who can help you safely stop study treatment. It may be dangerous to suddenly stop study treatment. The study doctor will also decide if you need to have any visits or tests to check on your health. If you withdraw from this study, you can still choose to be treated at MD Anderson.

If you stop being in the research, already collected data may not be removed from the study database. You may be asked whether the study doctor can continue to collect data from your routine medical care. If you agree, this data will be handled the same as research data.

- 6. This study or your participation in it may be changed or stopped without your consent at any time by the study chair, GlaxoSmithKline, Inc., the U.S. Food and Drug Administration (FDA), the Office for Human Research Protections (OHRP), or the IRB of MD Anderson. Possible reasons your participation in this study may be stopped include if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.
- 7. You will be informed of any new findings or information that might affect your willingness to continue taking part in the study and you may be asked to sign another informed consent and authorization form stating your continued willingness to participate in this study.

Most tests done on samples in research studies are only for research and have no clear meaning for health care. If the research with your identifiable information or samples gives results that do have meaning for your health, the researchers will not contact you to let you know what they have found.

- 8. MD Anderson may benefit from your participation and/or what is learned in this study.
- 9. This study is supported by: GlaxoSmithKline, Inc.
- 10. In a medical emergency, you may be cared for by someone who has a financial interest with the study sponsor(s)/supporter. If you have any questions about this, you may call the IRB at 713-792-6477.

#### **Future Research**

#### Data

Your personal information is being collected as part of this study. These data may be used by researchers at MD Anderson and GlaxoSmithKline, Inc. and/or shared with other researchers and/or institutions for use in future research.

#### Samples

Samples (such as blood and/or tissue) are being collected from you as part of this study. Researchers at MD Anderson may use any leftover samples that are stored at MD Anderson in future research. Leftover samples stored by GlaxoSmithKline, Inc. may be used in future research.

Before being used or shared for future research, every effort will be made to remove your identifying information from any data and/or research samples. If all identifying information is removed, you will not be asked for additional permission before future research is performed.

In some cases, all of your identifying information may not be removed before your data or research samples are used for future research. If future research is performed at MD Anderson, the researchers must get approval from the Institutional Review Board (IRB) of MD Anderson before your data and/or research samples can be used. At that time, the IRB will decide whether or not further permission from you is required. The IRB is a committee of doctors, researchers, and community members that is responsible for protecting study participants and making sure all research is safe and ethical.

If you do not want your samples or data to be used for future research, tell the study doctor. You may withdraw your samples at any time by telling your study team. If you decide to withdraw your samples, they will be returned to the lab they came from or destroyed. However, the data and test results already collected from your samples will be kept and may be used.

If this research is not performed at MD Anderson, MD Anderson will not have oversight of any data and/or samples.

#### Genetic Research

Research samples collected from you as part of this study may be used for genetic research, which may include whole genome sequencing. Whole genome sequencing is a type of testing in which researchers study your entire genetic makeup (DNA). This may help researchers learn how changes in the ordering of genes may affect a disease or response to treatment. If genetic research is done with your samples, those who have access to those samples may be able to identify you. The results of this research may also be able to be linked to you. The same level of data protection that covers your individual data does not apply to summary results (when data from the whole study is combined).

A federal law, called the Genetic Information Nondiscrimination Act (GINA), generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when deciding to hire, promote, or fire you or when setting the terms of your employment.

Be aware that this federal law does not protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance. Nor does this federal law prohibit discrimination based on an already known genetic disease or disorder.

#### **Outside Care**

Part of your care may be provided outside of MD Anderson by your home doctor(s).

### **Conflict of Interest**

Dr. Hans Lee (Co-PI) has received compensation from GlaxoSmithKline as a Consultant. The financial interests are within the limits of the conflict of interest policy.

Dr. Nimisha Patel (Collaborator) has received compensation for providing services to GSK Biologicals. The financial interests are within the limits of the conflict of interest policy.

# <u>Authorization for Use and Disclosure of Protected Health Information (PHI):</u>

- A. During the course of this study, MD Anderson will be collecting and using your PHI, including identifying information, information from your medical record, and study results. For legal, ethical, research, and safety-related reasons, your doctor and the research team may share your PHI with:
  - Federal agencies that require reporting of clinical study data (such as the FDA, National Cancer Institute [NCI], and OHRP)
  - The IRB and officials of MD Anderson
  - GlaxoSmithKline, Inc., who is a supporter of this study, and/or any future sponsors/supporters of the study
  - Study monitors and auditors who verify the accuracy of the information
  - Individuals who put all the study information together in report form

Study sponsors and/or supporters receive limited amounts of PHI. They may also view additional PHI in study records during the monitoring process. MD Anderson's contracts require sponsors/supporters to protect this information and limit how they may use it.

To protect your identity, the samples collected from you will be labeled a unique number instead of your name or other identifying information. Only the study doctor or study staff will have access to the code that can link you to your samples.

The results of this research may be published in scientific journals or presented at medical meetings, but your identity will not be disclosed.

- B. Signing this consent and authorization form is optional but you cannot take part in this study or receive study-related treatment if you do not agree and sign.
- C. MD Anderson will keep your PHI confidential when possible (according to state and federal law). However, in some situations, the FDA could be required to reveal the names of participants.

- Once disclosed outside of MD Anderson, federal privacy laws may no longer protect your PHI.
- D. The permission to use your PHI will continue indefinitely unless you withdraw your authorization in writing. Instructions on how to do this can be found in the MD Anderson Notice of Privacy Practices (NPP) or you may contact the Chief Privacy Officer at 713-745-6636. If you withdraw your authorization, you will be removed from the study and the data collected about you up to that point can be used and included in data analysis. However, no further information about you will be collected.
- E. A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### **CONSENT/AUTHORIZATION**

I understand the information in this consent form. I have had a chance to read the consent form for this study, or have had it read to me. I have had a chance to think

about it, ask questions, and talk about it with others as needed. I give the study chair permission to enroll me on this study. By signing this consent form, I am not giving up any of my legal rights. I will be given a signed copy of this consent document. SIGNATURE OF PARTICIPANT DATE PRINTED NAME OF PARTICIPANT WITNESS TO CONSENT I was present during the explanation of the research to be performed under this protocol. SIGNATURE OF WITNESS TO THE VERBAL CONSENT DATE PRESENTATION (OTHER THAN PHYSICIAN OR STUDY CHAIR) A witness signature is only required for non-English speakers utilizing the short form consent process (VTPS) and patients who are illiterate. PRINTED NAME OF WITNESS TO THE VERBAL CONSENT PERSON OBTAINING CONSENT I have discussed this research study with the participant and/or his or her authorized representative, using language that is understandable and appropriate. I believe that I have fully informed this participant of the nature of this study and its possible benefits and risks and that the participant understood this explanation. PERSON OBTAINING CONSENT DATE

PRINTED NAME OF PERSON OBTAINING CONSENT